CLINICAL TRIAL: NCT01935687
Title: Clinical Evaluation of Instrumented Wheel of Wheelchair as Biomedical Device Quantifying the Displacement Efficiency
Brief Title: Clinical Evaluation of Instrumented Wheel as Biomedical Device Quantifying the Displacement Efficiency
Acronym: FRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P101006
Record Dates: First submitted 2013-03-04; First posted 2013-09-05 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Spinal Cord Injury
Keywords: Instrumented Wheel; Manual Wheelchair; Spinal Cord Injury (SCI); Manual wheelchair Users; Aged between 18-70 years
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Using of instrumented wheel and ergometer roller (Experimental): The same patient will receive two types of tests: instrumented wheel and ergometer roller.
  Interventions: Device: Using of instrumented wheel; Device: Using of ergometer roller

INTERVENTIONS:
Device: Using of instrumented wheel — Using of instrumented wheel
Device: Using of ergometer roller — Using of ergometer roller

SUMMARY:
The purpose of this study is to validate an instrumented wheel such as a new biomedical device. The physicians will compare this instrumented wheel with another instrumentation "Ergometer roller", each patient will try the both instrumentations, physical and physiological parameters will be measured.

The increase rate of radial power during the cardiac stress test may be more important when the physicians use the instrumented wheel.

DETAILED DESCRIPTION:
* The manual wheelchair is used by people for whom walking is difficult or impossible due to spinal cord lesions, neurological and muscular diseases, lower limb trauma, age …etc.

Although the wheelchair help to regain mobility, this made of displacement is nor natural nor well-to-do.

* The CIC-IT and TSR (Transmissions Services Roulements, Mérignac, France) improved the instrumented wheel, adaptable with all wheelchairs, with information wireless transmission.
* The primary objective of study is to validate the instrumented wheel of manual wheelchair such as a new device of evaluation of capacities of displacement in ecologic situation.
* The primary criteria is to compare the mechanical power calculated using instrumented wheel versus the power calculated using ergometer roller during protocol of standard cardio-respiratory stress test.

This study is interventional, mono-centric, controlled and crossover. The population concerned is patients with spinal cord injury (SCI) and users of manual wheelchair.

Number of subjects projected for the entire study: 62 patients The total duration of participation of each patient: 7 days ±2days

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-70 years.
* Spinal cord injured patient.
* User of manual wheelchair for daily locomotion (having at least 30/100 at displacement items of WST questionnaire) .
* Affiliation to a social security scheme or entitled.
* Informed consent dated and signed by subject or subject's legally acceptable representative (and investigator).

Exclusion Criteria:

* Cognitive troubles.
* Progressive diseases: Tumoral, infectious, inflammatory and associated pathologies: brain injury, amputation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Mechanical power calculated by instrumented wheel and ergometer roller. | 20 min
  Comparison between mechanical power calculated by the instrumented wheel and mechanical power calculated by ergometer roller.

SECONDARY OUTCOMES:
Efficient fraction of total power calculated using instrumented wheel | 6 min
  Tangential power / total power
Efficient fraction of total power calculated using ergometer roller | 15 min
  Tangential power / total power

OTHER OUTCOMES:
Physiological parameters using instrumented wheel | 6 min
  Heart rate, VO2 and Borg score.
Physiological parameters using ergometer roller | 15 min
  Heart rate, VO2 and Borg score.

CONTACTS AND LOCATIONS:
Overall Officials: Djamel Bensmail, MD, Principal Investigator — Physical medicine and rehabilation Department, Hôpital RAYMOND POINCARE, 92380 Garches, France
Locations (1):
- Djamel Bensmail, Garches, Hauts-de-Seine, France